CLINICAL TRIAL: NCT03384095
Title: Single Center, Placebo-Controlled Trial of Oral High-Molecular Weight Hyaluronic Acid for the Prevention of Aromatase Inhibitor-Associated Arthralgias
Brief Title: Trial of Oral Hyaluronic Acid for the Prevention of Aromatase Inhibitor-Associated Arthralgias
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study abandoned prior to opening to accrual or study start
Sponsor: Erin Newton (Other)
Collaborators: Indiana University (Other); NOW Foods (Other)
Responsible Party: Sponsor-Investigator, Erin Newton, Assistant Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IUSCC-0533
Record Dates: First submitted 2017-12-18; First posted 2017-12-27 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Breast Neoplasm Female; Arthralgia
Keywords: Aromatase Inhibitors
MeSH Terms: conditions — Arthralgia | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid (Experimental): Subjects in this arm will be given 100 mg of hyaluronic acid in capsule form. Subject in this arm will be asked to 1 capsule take twice daily for 26 weeks.
  Interventions: Drug: Hyaluronic Acid (HA)
- Placebo (Placebo Comparator): Subjects in this arm will be given a placebo comparator capsule that is identical to the hyaluronic capsule containing microcrystalline cellulose as the sole ingredient. Subjects in this arm will be asked to take 1 capsule twice daily for 26 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hyaluronic Acid (HA) — Dosage form: hyaluronic capsules; Dose: 100 mg; Frequency: twice daily; Duration: 26 weeks
  Arms: Hyaluronic Acid
Other: Placebo — Dosage form: microcrystalline cellulose (MCC) capsules; Dose: approx. 100 mg (determined by weight of HA counterpart); Frequency: twice daily; Duration: 26 weeks
  Arms: Placebo

SUMMARY:
This is a single center, double-blinded, placebo-controlled, randomized Phase II trial to determine whether oral hyaluronic acid will prevent aromatase inhibitor (AI)-associated arthralgias. Subjects must have ER/PR-positive breast cancer tumor with history of aromatase inhibitor-associated musculoskeletal symptoms (AIMSS) which resolved after cessation of their AI (anastrazole or letrozole) within 90 days of enrollment. Subjects will be stratified by initial AI, thus within each initial AI, subjects will be randomized to receive either the experimental treatment (hyaluronic acid) or placebo. Subjects will begin the assigned treatment for 2 weeks prior to transitioning to the second AI. Evaluations will be taken at baseline, 6 weeks (1 month on study drug and AI), 14 weeks (3 months on study drug and AI), and at 26 weeks (6 months on study drug and AI). Treatment with hyaluronic acid and placebo will last for 26 weeks total.

DETAILED DESCRIPTION:
Primary Objective To determine whether oral HA will prevent AI-induced arthralgias and preserve physical function.

Secondary Objectives

1. To explore whether oral HA will have an acceptable safety and tolerability profile.
2. To determine whether oral HA will prevent other AI associated symptoms as assessed by patient reported outcomes (PRO's).
3. To assess how many of the subjects are 90% compliant with taking the HA as directed.

Exploratory Objective To determine if mi486, (a microRNA enriched in skeletal muscle) and other biomarkers associated with AIMSS (TNF, IL-6, IL-17) vary with the administration of HA.

ELIGIBILITY:
Study Population ER/PR-Positive Breast Cancer Subjects whose AIMSS resolved with cessation of their AI and are candidates for switching to a different AI and who meet the inclusion and exclusion criteria will be eligible for participation in this study.

Inclusion Criteria

1. Age ≥ 18 years old.
2. Had been taking anastrazole or letrozole, and discontinued it within the past 90 days due to pain and/or stiffness. The AI-related pain/stiffness must have resolved.
3. Prior tamoxifen use is allowed.
4. A prior switch from exemestane is allowed.
5. Women who have undergone a total mastectomy or breast conserving surgery for Stage 0-3 breast cancer +/- chemotherapy, +/- antiHer2Neu therapy, +/- radiotherapy.
6. Must have ER and/or PR positive tumors.
7. Women who are postmenopausal by the presence of natural amenorrhea ≥ 12 months or by ovarian ablation (bilateral oophorectomy, radiation, or administration of a gonadotropin-releasing hormone agonist).
8. Eastern Cooperative Oncology Group Performance Score (ECOG PS) 0-3 (Appendix II).
9. Patients may or may not be taking non-opioid analgesics.
10. Adequate renal and hepatic function:

    i) Include only subjects with AST and ALT < 2.0 × ULN; AP < 1.5 × ULN; total bilirubin < 1.2 × ULN ii) Include only subjects with as calculated creatinine clearance (CrCl) > 60 mL/min determined by the central laboratory using the modified Cockcroft-Gault equation; blood urea nitrogen (BUN) < 1.5 × upper limit of normal (ULN)
11. Written informed consent from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria

1. Presence of residual or recurrent cancer.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Consumption of HA-containing supplements in the four weeks prior to study.
4. Known allergy to microcrystalline cellulose or HA. Any questionable reaction to injected HA will be thoroughly investigated.
5. Prolonged systemic corticosteroid treatment, except for topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airway diseases), eye drops or local insertion (i.e., intra-articular). A short duration of systemic corticosteroids is allowed but not within 30 days prior to registration.
6. Self-reported compliance issues and lack of regular prescription filling.
7. Previous diagnosis of fibromyalgia and/or rheumatoid arthritis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Difference in mean change in joint pain between HA and placebo groups | 14 weeks
  As measured by the Brief Pain Inventory - Short Form (BPI-SF) questions #3-#6, #9A-G. This 14-item questionnaire was developed for use in patients with cancer that uses a scale from 0 to 10 to assess worst pain, pain severity, and pain interference over the past week. The first 8 items have to do with the severity of the pain, and the remaining 7 items ask about how the pain has affected function.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (i.e. safety and tolerability of HA) | 30 weeks
  Summary of adverse events as measured by CTCAE v4.0
Difference in mean joint symptoms between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) scores. This questionnaire assesses the three domains of pain, stiffness, and physical function in the lower extremities over the past 7 days. It is scored from 0 to 100, with higher scores indicating worse symptoms.
Difference in mean joint function between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Disabilities of the Arm, Shoulder, and Hand questionnaire (QuickDASH) scores. This 11-item instrument assesses physical function and symptoms in patients with musculoskeletal disorders of the upper limbs. It is a questionnaire scored from 1 to 5, with the higher score indicating worse symptoms, and there is a validated method to calculate a single Disability/Symptom Score.
Difference in mean quality of sleep between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Pittsburgh Sleep Quality Index (PSQI) scores. This an 18-item instrument produces a global sleep-quality score and the following component scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction.
Difference in global change between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Patient's Global Impression of Change scale (PGIC) scores
Difference in mean change in WOMAC subscale 1 scores between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) subscale 1 scores. As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) scores. This questionnaire assesses the three domains of pain, stiffness, and physical function in the lower extremities over the past 7 days. It is scored from 0 to 100, with higher scores indicating worse symptoms.
Difference in mean change in WOMAC subscale 2 scores between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) subscale 2 scores. As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) scores. This questionnaire assesses the three domains of pain, stiffness, and physical function in the lower extremities over the past 7 days. It is scored from 0 to 100, with higher scores indicating worse symptoms.
Difference in mean change in WOMAC subscale 3 scores between HA and placebo groups | 6, 14, and 26 weeks
  As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) subscale 3 scores. As measured by Western Ontario and McMaster osteoarthritis index (WOMAC) scores. This questionnaire assesses the three domains of pain, stiffness, and physical function in the lower extremities over the past 7 days. It is scored from 0 to 100, with higher scores indicating worse symptoms.
Time to discontinuation of second aromatase inhibitor due to AIMSS between HA and placebo groups | 26 weeks
  As measured by patient self-report of mediation compliance (medication diary) and chart review
Proportion of patients that remain on second aromatase inhibitor between HA and placebo groups | 26 weeks
  As measured by patient self-report of mediation compliance (medication diary) and chart review
Rate of 90% compliance between HA and placebo groups | 26 weeks
  As measured by patient self-report of mediation compliance (medication diary)
Mean frequency of as needed analgesia between HA and placebo groups | 6, 14, and 26 weeks
  As measured by patient self-report of mediation compliance (medication diary)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Newton, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts KE, Adsett IT, Rickett K, Conroy SM, Chatfield MD, Woodward NE. Systemic therapies for preventing or treating aromatase inhibitor-induced musculoskeletal symptoms in early breast cancer. Cochrane Database Syst Rev. 2022 Jan 10;1(1):CD013167. doi: 10.1002/14651858.CD013167.pub2. PMID 35005781